CLINICAL TRIAL: NCT02393261
Title: Validity and Security of 2500ml Huaren Peritoneal Dialysate: A Prospective, Randomized, Controlled, Multi-Center Clinical Trial
Brief Title: A Controlled and Multi-Center Study of 2500ml Huaren Peritoneal Dialysate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, The Sixth Affiliated Hospital of Sun Yat-Sen University, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Usix -2500PD-001
Record Dates: First submitted 2015-03-09; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Disorders Associated With Peritoneal Dialysis
MeSH Terms: interventions — Dialysis Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A 2500mlGroup (Experimental): use 2-3 bags of 2500ml Huaren dialysate in the daytime and keep 1 bag of 2500ml Huaren dialysate in the night
  Interventions: Other: 2500ml Huaren peritoneal dialysate
- B 2000mlGroup (Active Comparator): use 3-4 bags of normal 2000ml dialysate in the daytime and keep 1 bag of 2000ml dialysate in the night
  Interventions: Other: 2000ml peritoneal dialysate

INTERVENTIONS:
Other: 2500ml Huaren peritoneal dialysate — use 2-3 bags of 2500ml Huaren dialysate in the daytime and keep 1 bag of 2500ml Huaren dialysate in the night
  Arms: A 2500mlGroup
Other: 2000ml peritoneal dialysate — use 3-4 bags of normal 2000ml dialysate in the daytime and keep 1 bag of 2000ml dialysate in the night
  Arms: B 2000mlGroup

SUMMARY:
This prospective, randomized, controlled, multi-center clinical trial will evaluate the validity and security of 2500ml Huaren Peritoneal Dialysate compared with normal 2000ml peritoneal dialysate.

DETAILED DESCRIPTION:
Peritoneal dialysis (PD) is one of important way of renal replacement treatment worldwide. In China, about 40,000 patients suffered from end stage renal disease treated with PD, and most of them used imported dialysate, of which the price carried a great burden. Now, cheaper domestic dialysate is accessed to the ESRD patients in china, but the efficacy and safety of which are not fully clear. And according to researches from Hongkong, 6000ml of dialysate every day is able to. Thus, we presume 3 bags of 2500ml Huaren dialysate will satisfy the everyday need of an normal Asian. This will be a prospective, randomized, controlled, multi-center study. Patients in treatment group will use 2-3 bags of 2500ml Huaren dialysate in the daytime and keep 1 bag of 2500ml Huaren dialysate in the night, while those in control group will use 3-4 bags of normal 2000ml dialysate in the daytime and keep 1 bag of 2000ml dialysate in the night for 12 weeks. After followed-up for 12 weeks, the adequacy of PD, residual kidney function , peritoneum function and QOL of patients will be evaluated.

ELIGIBILITY:
Inclusion criteria:

1. The duration of PD is more than 1 month.
2. The age is range from 18 to 80 years old.
3. The patient can be treated with regular PD in home.
4. The volume of peritoneal dialysate is from 8L to 10 L in 1 day.
5. The patient can be visited regularly.
6. The patient must be freely given informed consent

Exclusion criteria:

1. Peritonitis was happened within 1 month
2. The KT/V<1.7
3. Infections in the exit or tunnel
4. With tumors.
5. With low transport of peritoneum.
6. With mental and behavior disorders.
7. With acute renal failure
8. Hemodialysis meanwhile
9. With heart failure( NYHA III-IV ) or cardio- cerebrovascular events
10. Attending other clinical trails
11. Refused to give informed consent Exit criteria

（1）Stop PD for more than 10 days （2）The patient demand to quit from the RCT （3）With serious adverse events.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-01; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Adequacy of dialysis (kt/v) | up to 8 weeks
  kt/v

SECONDARY OUTCOMES:
Residual kidney function (Residual kidney kt/v) | up to 6 months
  Residual kidney kt/v
Peritoneal function (Peritoneal equilibration test) | up to 6 months
  Peritoneal equilibration test

CONTACTS AND LOCATIONS:
Overall Officials: Zongpei Jiang, M.D. & Ph.D., Principal Investigator — The Sixth Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Nephrology, 6th Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China